CLINICAL TRIAL: NCT02250196
Title: A Randomized, Prospective Tiral on Efficacy and Tolerability of Low-volume Bowel Preparation Methods for Colonoscopy
Brief Title: A Randomized Prospective Trial Comparing Low-volume Bowel Preparation Methods
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, In-Kyung Yoo, fellow, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Korea University Prep
Record Dates: First submitted 2014-09-08; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Colorectal Cancer; Colon Adenoma
Keywords: Bowel preparation; Polyethylene glycol with ascorbic acid; Sodium picosulfate with magnesium citrate
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-Asc (Active Comparator): group 1 (PEG-Asc, N=100) received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure
  Interventions: Drug: PEG-Asc
- SPMC 2 (Active Comparator): group 2 (SPMC 2, N=100) received one sachet of SPMC at 7 p.m the evening before colonoscopy and another sachet of SPMC at 5 hours before procedure
  Interventions: Drug: SPMC 2

INTERVENTIONS:
Drug: PEG-Asc — received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure
  Other Names: Coolprep®; TaeJoon Pharmaceuticals, Seoul, Korea
  Arms: PEG-Asc
Drug: SPMC 2 — received one sachet of SPMC at 7 p.m the evening before colonoscopy and another sachet of SPMC at 5 hours before procedure
  Other Names: Picolight(Pharmbio korea, Seoul, Korea)
  Arms: SPMC 2

SUMMARY:
Colonoscopy is a common screening method to detect polyps and CRC. With the early detection of CRC through screening colonoscopy, patients could have better therapeutic effects and outcomes. In population screening programs, an increase in completed colonoscopies is related to a decrease in mortality from CRC. However, the miss rate for detecting colorectal neoplastic polyps of colonoscopy is 5-28%. The reluctance of participants to undergo bowel preparation results in the relatively low rate of detection of polyps and CRC, because poor preparation interferes with successful colon mucosa examination during a colonoscopy.

Low-volume bowel preparations provide equivalent cleansing effect compared with standard 4 liter polyethylene glycol. However, studies comparing the superiority between low-volume bowel preparations are rare, and results are controversial. This study aimed to compare the bowel cleansing quality and tolerability between split-dose sodium picosulfate/magnesium citrate and polyethylene glycol with ascorbic acid.

DETAILED DESCRIPTION:
1. Study design: endoscopist-blinded, prospective, randomized controlled trial
2. Subjects

   1. Entry criteria: Male or female patients, aged between18 and 80 years undergoing elective outpatient colonoscopy were eligible for the study.
   2. Exclusion criteria:

   patients who had chronic kidney disease, severe heart failure(New York Heart Association [NYHA] class III or IV), uncontrolled hypertension (systolic pressure ≥170 mm Hg, diastolic pressure ≥100 mm Hg), severe constipation, any bowel resection, significant gastroparesis, or suspected bowel obstruction or perforation.
3. Sampling design: Consecutive recruitment of consenting patients
4. Variables Predictor

   1. group 1 (SPMC 2) received one sachet of SPMC at 7 p.m the evening before colonoscopy and another sachet of SPMC at 5 hours before procedure
   2. group 2 (PEG-Asc) received 1 L solution of PEG-Asc at 7 p.m the evening before colonoscopy and another 1 L solution of PEG-Asc at 5 hours before procedure;
5. Primary Outcome: Quality of bowel preparation (Boston Bowel Preparation Scale, Aronchick scale, bubble score)
6. Secondary Outcome: Tolerability, palatability

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged between18 and 80 years undergoing elective outpatient colonoscopy were eligible for the study

Exclusion Criteria:

* patients who had chronic kidney disease, severe heart failure(New York Heart Association [NYHA] class III or IV), uncontrolled hypertension (systolic pressure ≥170 mm Hg, diastolic pressure ≥100 mm Hg), severe constipation, any bowel resection, significant gastroparesis, or suspected bowel obstruction or perforation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
the quality of the bowel preparation using Preparation Scale | 20 minutes
  Preparation Scale

SECONDARY OUTCOMES:
Completeness of the bowel preparation | 30 minutes before the colonoscopy
  Patient compliance was recorded by checking the completeness of the prescribed preparation methods including bowel cleansing agent solution and recommended clear liquid.
the patient's tolerability | 30 minutes before the colonoscopy
  Patients were asked with questionnaires about the symptoms associated with the preparation to assess the patients' tolerability before the colonoscopy. Patients were asked whether they experienced any of the following : abdominal fullness, cramping, nausea, vomiting, sleep disturbance, and overall discomfort, and these symptoms were scored on a 5-point scale where 1 = "none", 2 = "mild", 3 = "moderate", 4 = "severe", and 5 = "very severe".

CONTACTS AND LOCATIONS:
Overall Officials: Eun Sun Kim, PhD, Study Director — Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, Republic of Korea; In Kyung Yoo, MD, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Korea University College of Medicine, Seoul, Republic of Korea
Locations (1):
- Korea University Anam Hospital, Seoul, Anamdong 5-ga, Seongbuk-gu, South Korea